CLINICAL TRIAL: NCT02466074
Title: Augmenting Cerebral Blood Flow to Treat Established Multiple Sclerosis
Acronym: perfuseMS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inadequate recruitment; termination of funding
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, John A. Lincoln, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC-MS-14-0450
Record Dates: First submitted 2015-06-03; First posted 2015-06-09 (Estimated); Results first posted 2023-03-01 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-03

CONDITIONS: Multiple Sclerosis
Keywords: Acetazolamide; Lesions; Neurodegeneration; Repair
MeSH Terms: conditions — Multiple Sclerosis; Nerve Degeneration | interventions — Acetazolamide

STUDY DESIGN:
Intervention Model Description: Two phase design: phase 1, patients randomized to ACZ or placebo and followed for 24 weeks; phase 2, patients that received placebo in phase 1 switch to ACZ (delayed-start group) and patients that received ACZ in phase 1 continue on ACZ (ACZ-ACZ group)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Acetazolamide (Experimental): Acetazolamide in oral daily divided dose administered for 6 consecutive months
  Interventions: Drug: Acetazolamide
- Placebo (Placebo Comparator): Placebo in oral daily divided dose administered for 6 consecutive months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetazolamide — see arm description
  Other Names: Diamox
  Arms: Acetazolamide
Drug: Placebo — Placebo arm
  Arms: Placebo

SUMMARY:
This study will evaluate how improved cerebral blood flow affects the way in which newly formed MS lesions evolve and whether tissue repair is improved. Patients with multiple sclerosis (MS) will be treated with acetazolamide in daily divided doses and obtain MRI to determine how much and in which regions of the brain cerebral perfusion improves as well as the extent to which tissue integrity is improved in these areas.

DETAILED DESCRIPTION:
Cerebral perfusion is altered in many disease states, including MS. Altered perfusion has been seen in patients with all multiple sclerosis (MS) phenotypes and is well established as occurring early in relapsing-remitting disease.

Previous research in our laboratory has shown that reduced cerebral perfusion in MS patients is a precursor to the formation of chronic lesions. In addition, studies have suggested that "virtual hypoxia", resultant from the combination of diminished cerebral perfusion and increased energy demand, contributes to tissue damage that strongly correlates with clinical disability in persons with MS. Our preliminary studies have already shown short-term increases in global and regional cerebral perfusion in MS patients after therapy with acetazolamide (ACZ).

The central hypothesis is that if cerebral perfusion is important in tissue injury, then MS lesions within hypoperfused areas are more likely to develop permanent tissue damage, and medications that improve cerebral perfusion might beneficially alter the evolution of MS plaques, enhance remyelination and repair and diminish clinical disability progression.

Sixty MS patients will be enrolled in this single-center exploratory RCT. Half of the patients will be randomly assigned to get ACZ treatment in phase 1 consisting of 24 weeks on ACZ, followed by another 24 weeks on ACZ during phase 2. The other half of the patients will be assigned to placebo for 24 weeks in phase 1 and then switched to ACZ and followed for 24 weeks in phase 2. This study will utilize various imaging techniques to determine the degree to which cerebral blood flow is improved in MS subjects after administration of ACZ.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of relapsing forms of multiple sclerosis using revised McDonald criteria
2. Stable on any FDA-approved disease-modifying therapy. The term "stable" implies that the subject has not had change in therapy for any reason for the 6 months prior to study entry.
3. Expanded Disability Status Scale (EDSS) score of 0-6.0 inclusive
4. Understood and signed written informed consent, obtained prior to the study subject undergoing any study related procedure, including screening tests.

Exclusion Criteria:

1. Known hypersensitivity to sulfonamides or derivatives
2. Known history of renal or hepatic disease, cerebrovascular disease including stroke, transient ischemic attack, myocardial infarction, angina or congestive heart failure.
3. Evidence to suggest hyponatremia or hypokalemia, marked kidney dysfunction defined as creatinine greater than 2.0 mg/dL or liver disease dysfunction defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) greater than three-fold upper limit of normal (ULN).
4. Evidence to suggest suprarenal gland failure.
5. Evidence of hyperchloremic acidosis.
6. Initiation of new immunosuppressant treatment after the subject becomes protocol-eligible (except for corticosteroids) or enrollment in a concurrent trial.
7. Prior treatment with mitoxantrone, natalizumab, methotrexate, cladribine cyclophosphamide or other change in disease modifying therapy (DMT) within 6 months of initiation of study.
8. Subjects with any history of cytopenia.
9. History of pulmonary obstruction or emphysema.
10. Active hepatitis B or hepatitis C infection or evidence of cirrhosis.
11. Human immunodeficiency virus (HIV) positivity.
12. Uncontrolled diabetes mellitus defined as HbA1c>8% and/or requiring intensive management.
13. Uncontrolled viral, fungal, or bacterial infection (excluding asymptomatic bacteriuria).
14. Any condition that, in the opinion of the investigators, would jeopardize the ability of the subject to tolerate treatment with ACZ.
15. Prior history of malignancy.
16. Positive pregnancy test or inability or unwillingness to use effective means of birth control. Effective birth control defines as:

    * Refraining from all acts of vaginal intercourse (abstinence)
    * Consistent use of birth control pills
    * Tubal sterilization or male partner who has undergone vasectomy
    * Placement of an intrauterine device (IUD)
    * Use, with every act of intercourse, of a diaphragm with contraceptive jelly and/or condoms with contraceptive foam
17. Presence of metallic objects implanted in the body that would preclude the ability of the subject to safely have MRI exams.
18. Psychiatric illness, mental deficiency, or cognitive dysfunction making compliance with treatment of informed consent impossible.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2016-08-17 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2022-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Lincoln, MD, PhD, Principal Investigator — UTHealth
Locations (1):
- UTHealth, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acetazolamide | Placebo
Started | 5 | 0
Completed | 5 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were assigned to the placebo arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Acetazolamide | Placebo | Total
Number analyzed (Participants) | 5 | 0 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (5.9) |  | 43.6 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 |  | 3
  Male | 2 |  | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 |  | 1
  Not Hispanic or Latino | 4 |  | 4
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 1 |  | 1
  White | 3 |  | 3
  More than one race | 0 |  | 0
  Unknown or Not Reported | 1 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 5 |  | 5

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Global Cerebral Blood Flow
Description: Percent change in global cerebral blood flow (CBF) after 24 weeks relative to pre-treatment baseline. Global CBF is determined using magnetic resonance imaging (MRI) methods.
  The data reported indicate the extent of change in global CBF--the higher the percent change, the greater the increase in global CBF and the better the outcome.
Time Frame: baseline, 24 weeks
Population: No participants were assigned to the placebo arm.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Acetazolamide | Placebo
Number analyzed (Participants) | 5 | 0
percent change | 22.9 (16.2) |

2. Secondary Outcome: Percent Change in Tissue Integrity in White Matter (Mean Diffusivity)
Description: The data reported indicate the extent of change in white matter integrity as determined using the diffusion tensor imaging-magnetic resonance imaging (DTI-MRI) measure of mean diffusivity. A positive percent change value indicates an increase in mean diffusivity between baseline and 24 weeks, and a higher mean diffusivity value indicates a breakdown in white matter integrity, so the greater the percent change, the greater the breakdown of white matter integrity and the worse the outcome.
Time Frame: baseline, 24 weeks
Population: No participants were assigned to the placebo arm.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Acetazolamide | Placebo
Number analyzed (Participants) | 5 | 0
percent change | 1.9 (1.3) |

3. Secondary Outcome: Percent Change in Tissue Integrity in White Matter (Fractional Anisotropy)
Description: The data reported indicate the extent of change in white matter integrity as determined using the diffusion tensor imaging-magnetic resonance imaging (DTI-MRI) measure of fractional anisotropy. A negative percent change value indicates a decrease in fractional anisotropy between baseline and 24 weeks, and a lower fractional anisotropy value indicates a breakdown in white matter integrity, so the lower (and more negative) the percent change, the greater the breakdown of white matter integrity and the worse the outcome.
Time Frame: baseline, 24 weeks
Population: No participants were assigned to the placebo arm.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Acetazolamide | Placebo
Number analyzed (Participants) | 5 | 0
percent change | -2.8 (2.4) |

4. Other Pre Specified Outcome: Composite Changes in Disability Measures
Description: Composite disability for an individual is defined as at least one of the following: a) any decrease in Expanded Disability Status Score (EDSS), b) 20% reduction in time to complete 9-Hole Peg Test (9HPT) for either the dominant or non-dominant hand, c) 20% decrease in Timed 25-Foot Walk (T25FW) or d) a >= 4-point or 10% improvement in accuracy for Symbol Digit Modalities Test (SDMT).
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: No participants were assigned to the placebo arm.
Arm/Group | Acetazolamide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/0
Other Adverse Events (participants affected / at risk) | 0/5 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-27): https://cdn.clinicaltrials.gov/large-docs/74/NCT02466074/Prot_SAP_000.pdf